CLINICAL TRIAL: NCT01743573
Title: Effects on Physical Fitness, Immunity, and Quality of Life of Yoga Training in Breast Cancer Survivors.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200811002R
Record Dates: First submitted 2012-11-20; First posted 2012-12-06 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- yoga training (Experimental): Yoga training
  Interventions: Other: yoga
- control (No Intervention): no yoga training

INTERVENTIONS:
Other: yoga
  Arms: yoga training

SUMMARY:
This study wants to prove that Yoga Training can improve physical Fitness, immunity, and quality of Life of in Breast Cancer Survivors. In summary, our findings show potential benefits of yoga for people with cancer in improvements of psychological health. Because of the small number of studies having been conducted and the methodological limitations, the results should be regarded as preliminary and treated with caution. Our preliminary findings also provide practitioners with important information that yoga may be a possible adjunctive therapy for cancer patients to help manage psychological distress and to improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer with stage1 or stage2, Sedentary life style, no orthopaedic disease and medical disease

Exclusion criteria

* recurrent or metastasis, medical or current psychiatric illness which would make compliance with the study protocol difficult or dangerous, medications which would alter training response

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
change from baseline immunological factors, cardiorespiratory and muscle fitness, questionnaire for physical activity, fatigue and quality of life at 13th weeks | 13th week

SECONDARY OUTCOMES:
change from baseline immunological factors, cardiorespiratory and muscle fitness, questionnaire for physical activity, fatigue and quality of life at 25th weeks | 25th week

CONTACTS AND LOCATIONS:
Overall Officials: Jau-Yih Tsauo, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan